CLINICAL TRIAL: NCT03035435
Title: Fast-track Rehabilitation After Total Knee or Hip Arthroplasty: an Observational Prospective Case-control Study
Brief Title: Fast-track Rehabilitation After Total Knee or Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Chiara Arienti, PhD, Fondazione Don Carlo Gnocchi Onlus
Other Study IDs: Fast Track Rehab
Record Dates: First submitted 2017-01-17; First posted 2017-01-30 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Knee Arthroplasty; Hip Arthroplasty
Keywords: fast-track rehabilitation; fast-track surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- study group: fast-track rehabilitation
  Interventions: Other: fast-track rehabilitation
- control group: standard care rehabilitation
  Interventions: Other: standard care rehabilitation

INTERVENTIONS:
Other: fast-track rehabilitation
  Groups: study group
Other: standard care rehabilitation
  Groups: control group

SUMMARY:
In the last years, a lot of surgical fast track programs (SFTP) have been created and developed. This is due to the steady growing number of interventions on knee and hip; after the surgical treatment, a period of physical rehabilitation (PR) is established to be useful and effective, it usually takes 2-3 weeks. The recovery of strength, range of motion (ROM), independence, the reduction of pain and disability are the aims of PR. With the SFTP and a specific rehabilitation program named fast track rehabilitation (FTR) these times can be reduced. First of all because the length of stay (LOS) it's also caused by organizational problems of the hospitals, not only for the factors related to the patient. It's already been demonstrated that an early mobilization decreases the risk of thromboembolic complications and of pain, furthermore an early rehabilitation increase the patient autonomy and reduces the lost of residual abilities. Moreover a PR program studied for fast track patient will reduce minimum by a 50% the LOS in hospital, decreasing so the sanitary efforts that are always a problem for all the countries. The aim of this study is therefore to propose a fast track rehabilitation program based on an 8 days program for hip and knee arthroplasty being operated with an SFTP.

ELIGIBILITY:
Inclusion Criteria:

* adult people (>18 years), both sex, admitted for elective total knee or hip arthroplasty, with a clinical stability (Hb>9 g/l).

Exclusion Criteria:

* the presence of pain measured with NRS (NRS>4)
* rheumatoid arthritis, past surgery
* cancer
* neurological and psychiatric disorders
* dementia with Minimental Test<24
* pregnancy
* participation in the other clinical studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The recruitment will take place to Rehabilitation Unit of Don Gnocchi Foundation of Rovato (Brescia, Italy), from January 2016 to August 2016. An informed consent will be signed by each participant in agreement with Helsinki Declaration. The study is approved by the local Ethical Committee.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
International Knee Society Score | Change from Baseline fast-track rehabilitation at 8th and 15th day
Merle D'Aubigne' scale | Change from Baseline fast-track rehabilitation at 8th and 15th day

SECONDARY OUTCOMES:
Barthel Index | Change from Baseline fast-track rehabilitation at 8th and 15th day

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Arienti, PhD(s), Principal Investigator — IRCCS Don Gnocchi Foundation